CLINICAL TRIAL: NCT04979559
Title: Development Mobile Health Application of Screening and Early Intervention for Prediabetic Patient at Primary Health Cares Setting: Protocol of a Pilot Study
Brief Title: Mobile Health Application of Screening and Early Intervention for Prediabetic Patient at Primary Health Cares Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Collaborators: Universitas Islam Indonesia (Other)
Responsible Party: Principal Investigator, Yaltafit Abror Jeem, Principle investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: KE/FK/1375/EC/2020
Record Dates: First submitted 2021-06-20; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: PreDiabetes; Prediabetic State
Keywords: Telemedicine; Intervention; Screening; Self Care; Primary Health Care
MeSH Terms: conditions — Prediabetic State | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two arms: (1) a group that is used mobile health application intervention for screening and early intervention and (2) a group that receive standard care for screening and early intervention from PHCs regular practice.
Who Masked: Participant, Care Provider
Masking Description: The participant and care provider in each site are unaware of the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth apps (Experimental): The participants in this arm will receive information regarding mobile health applications used for screening and early intervention of the prediabetic states.
  Interventions: Device: Mobile health apps
- Standard care (Active Comparator): The participant in this arm will receive regular practice or standard care of screening and early intervention of prediabetic state.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Mobile health apps — Mobile health application intervention including screening and early intervention such as diet and physical activity suggestion
  Arms: mHealth apps
Other: Standard care — Regular practice for screening and early intervention for prediabetes patient in primary health cares setting
  Arms: Standard care

SUMMARY:
Background: Preventing type-2 diabetes mellitus begins with early screening and intervention of prediabetic participants. Until now, prediabetes screening and early intervention have not been optimal. The rapid advancement of technology, as well as its increased use, may provide an opportunity to improve the quality and cost of healthcare services. It is quite practicable to investigate and implement a valid, practical and easy-to-use mobile health application for participants and health staffs in screening and early intervention of prediabetes participants at primary health cares setting. This protocol aimed to identify and develop a valid, practical, and easy-to-use mobile health application for screening and early intervention of prediabetes participants at primary health cares.

Methods: This protocol was prepared in accordance with the Standard Protocol Items: Recommendations for Interventional Trials 2013 statement. This is a mixed-methods study with sequential exploratory approach. This project will begin with in-depth interview to gather qualitative information regarding mobile health application necessity for prediabetes participants at the primary health cares. The impact of the usage will be studied quantitatively using randomized controlled trial. Prediabetic participants and primary health cares staffs at Yogyakarta province will be the research subjects. The collected findings will be examined based on the type of the data.

Discussion: The proposed research aimed to obtain information and trial results regarding mobile health application usage for prediabetes participants screening and early intervention at primary health cares setting.

DETAILED DESCRIPTION:
The goal of this study is to create a mobile health application for prediabetes patients that included screening and early intervention in Primary Health Cares (PHCs) setting. More specifically, the objectives are as follows:

1. To portray regular prediabetes screening and early intervention practice in PHCs.
2. To assess prediabetes screening and early intervention data necessity for mobile health application model at PHCs.
3. To assess the feasibility of mobile health application usage for screening and early intervention of prediabetes patients at PHCs.
4. To assess internal and external factors that influence the intention-to-use, easiness, and usefulness of mobile health applications for prediabetes patients and health staff.
5. To assess the impact of early intervention using mobile health applications on prediabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as the prediabetic state using American Diabetes Association (ADA) criteria
* have no previous diagnosis of type 2 diabetes or history of taking anti-hyperglycemic drugs
* have access to and able to use a personal smartphone
* willing to undertake study activities and written informed consent

Exclusion Criteria:

* severe medical condition
* disability to perform physical activity

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Body weight mean change from baseline | at baseline and after intervention at 12-weeks
  Participants' body weight measured by scales using kilograms (kg) measurement unit
Waist circumference mean change from baseline | at baseline and after intervention at 12-weeks
  Participants' waist circumference measured using measuring tape in centimeter (cm) measurement unit
Fasting blood glucose mean change from baseline | at baseline and after intervention at 12-weeks
  Participants' fasting blood glucose measured from vein blood in milligram per deciliter (mg/dL) measurement unit
Hemoglobin A1c mean change from baseline | at baseline and after intervention at 12-weeks
  Participants' Hemoglobin A1c measured from vein blood in percent
Oral glucose tolerance test mean change from baseline | at baseline and after intervention at 12-weeks
  Participants' oral glucose tolerance test measured from vein blood in milligram per deciliter (mg/dL) measurement unit

SECONDARY OUTCOMES:
Area under the curve of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  screening accuracy of the instrument reported using graph
Sensitivity value of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Sensitivity value of the instrument calculated using formula derived from 2x2 tables of diagnostic test
Specificity value of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Specificity value of the instrument calculated using formula derived from 2x2 tables of diagnostic test
Positive predictive value of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Positive predictive value of the instrument calculated using formula derived from 2x2 tables of diagnostic test
Negative predictive value of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Negative predictive value of the instrument calculated using formula derived from 2x2 tables of diagnostic test
Accuracy value of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Accuracy predictive value of the instrument calculated using formula derived from 2x2 tables of diagnostic test
Likelihood ratio of screening instrument compared to American Diabetes Association criteria | immediately after the intervention begin
  Likelihood ratio of the instrument calculated using formula derived from 2x2 tables of diagnostic test

OTHER OUTCOMES:
Participant's acceptance of mobile health application | after intervention at 12-weeks
  evaluation of participant's acceptance to the device using Mobile Health Application Acceptance Questioner adapted from previous study

CONTACTS AND LOCATIONS:
Overall Officials: Yaltafit A Jeem, Principal Investigator — Gadjah Mada University
Locations (1):
- Kalasan PHC, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No